CLINICAL TRIAL: NCT00182585
Title: Computer-Assisted HIV Prevention for Young Drug Users
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Development and Research Institutes, Inc. (Other)
Collaborators: Daytop (adolescent treament program) (Unknown); St. Luke's-Roosevelt Hospital Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA015964 (NIH)
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2008-08-13 (Estimated); Status verified 2008-08

CONDITIONS: HIV
Keywords: HIV; hepatitis; STDs; adolescents; addiction; treatment; prevention; HIV and related risk behavior among youth in drug treatment
MeSH Terms: conditions — Hepatitis; Sexually Transmitted Diseases; Behavior, Addictive

INTERVENTIONS:
Procedure: computer-based HIV, STD & Hepatitis Education
Procedure: educator-delivered HIV, STD and Hepatitis education

SUMMARY:
In this study, the investigators are developing and evaluating an interactive, computer-assisted HIV, STD and disease prevention program for young substance abusers that incorporates effective components of both prevention science and educational technologies.

DETAILED DESCRIPTION:
Adolescents and young adults who use drugs are at high risk for infection with HIV, STDs and other diseases with similar transmission dynamics. Although several age-appropriate and effective HIV, STD and disease prevention efforts have been identified for young substance abusers, most interventions have been narrow in focus and are generally not structured to readily address changing patterns of drug use among adolescents that place them at risk for infection with these diseases. In this study, we are developing and evaluating an interactive, computer-assisted HIV, STD and disease prevention program for young substance abusers that incorporates effective components of both prevention science and educational technologies. We plan to develop this program with the input from the target population of adolescents and young adults. We also plan to conduct a randomized, controlled trial to evaluate the benefit of including this program in HIV and disease prevention efforts with youth in substance abuse treatment. In so doing, we will evaluate the ability of the program to promote accurate knowledge about HIV and other diseases, promote self-efficacy to reduce risk behavior and change actual rates of risk behavior among young substance abusers. This computer-based program will be designed to promote the increased adoption of effective HIV and disease prevention science for this population. New information about changing patterns of drug use and HIV risk behaviors can be readily incorporated into the program as it becomes available. The program can be easily exported and able to be applied with fidelity. Importantly, the program will be structured such that a therapist or educator may customize the program content for use by various sub-populations of substance-abusing adolescents and young adults. Thus, the program will be able to address risk factors specific to each young drug user. This program may address many of the challenges associated with the current delivery of evidence-based HIV prevention programs to this population.

ELIGIBILITY:
Inclusion Criteria:

* Aadolescents in outpatients substance abuse treatment
* Ages 13 - 18 years
* Within first month of treatment entry

Exclusion Criteria:

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2004-08

PRIMARY OUTCOMES:
HIV risk behavior

SECONDARY OUTCOMES:
knowledge related to HIV, Hepatitis, STDs
behavioral intentions
attitudes toward risk-reduction behavior
feedback on intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marsch, PhD, Principal Investigator — National Development and Research Institutes, Inc.
Locations (2):
- United States (2):
  - Daytop, Brooklyn, New York
  - St. Luke's-Hospital, CAPA Program, New York, New York